CLINICAL TRIAL: NCT00482053
Title: A Phase 2 Study in Poor Risk Diffuse Large B-cell Lymphoma of Total Lymphoid Irradiation & Antithymocyte Globulin Followed by Matched Allogeneic Hematopoietic Transplantation as Consolidation to Autologous Hematopoietic Cell Transplantation
Brief Title: Phase 2 Poor Risk DLBCL of TLI and ATG Followed by Matched Allogeneic HT as Consolidation to Autologous HCT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Wen-Kai Weng, Assistant Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-06703; 97355 (Other: Stanford University alternate IRB Number); BMT186 (Other: OnCore number)
Record Dates: First submitted 2007-05-31; First posted 2007-06-04 (Estimated); Results first posted 2018-05-14 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Lymphoma, B-cell; Lymphoma, Non-Hodgkin; Diffuse Large B-cell Lymphoma (DLBCL); Malignant Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse | interventions — Transplantation; Rituximab; Carmustine; Etoposide; etoposide phosphate; Filgrastim; Granulocyte Colony-Stimulating Factor; Antilymphocyte Serum; Cyclosporine; Mycophenolic Acid; Cyclophosphamide; Acetaminophen; Diphenhydramine; Hydrocortisone; Methylprednisolone; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Auto-HCT followed by Allo-HCT for Poor-risk DLBCL (Experimental): Participants will have peripheral blood stem cells (PBSC, aka progenitor / stem cells) mobilized to peripheral blood with rituximab, chemotherapy (cyclophosphamide or etoposide), and filgrastim; undergo apheresis to collect (self/autologous PBSC), and receive carmustine, etoposide, and cyclophosphamide as conditioning for PBSC infusion as a hematopoietic cell transplant (auto-HCT).
  Then participants will receive allogeneic HCT (allo-HCT) transplant conditioning [total lymphoid irradiation (TLI) + anti-thymocyte globulin (ATG)] followed by allogenic PBSC (allo-HCT) obtained from a human leukocyte antigen (HLA)-matched or single mismatch filgrastim-mobilized donor. Participant allo-HCT transplant is to occur within 150 days of auto-HCT. Post-allo-HCT treatment includes cyclosporine + mycophenolate mofetil (MMF).
  Subject's participation ends if donor is not identified within 150 days. Pre-medication includes acetaminophen; diphenhydramine; hydrocortisone; & methylprednisolone.
  Interventions: Procedure: Autologous hematopoietic stem cell transplantation (auto-HSCT); Procedure: Allogeneic hematopoietic stem cell transplantation (allo-HSCT); Procedure: Total lymphoid irradiation (TLI); Drug: Rituximab; Drug: Carmustine; Drug: Etoposide; Drug: Filgrastim; Drug: Anti-thymocyte globulin (ATG); Drug: Cyclosporine; Drug: Mycophenolate mofetil (MMF); Drug: Cyclophosphamide; Drug: Acetaminophen; Drug: Diphenhydramine; Drug: Hydrocortisone; Drug: Methylprednisolone

INTERVENTIONS:
Procedure: Autologous hematopoietic stem cell transplantation (auto-HSCT) — Auto-HCT involves an intravenous infusion of a participant's previously collected and frozen white blood cells collected after treatment with mobilizing agents
  Other Names: Autologous peripheral blood progenitor cell (PBPC) transplantation
Procedure: Allogeneic hematopoietic stem cell transplantation (allo-HSCT) — Allo-HCT involves an intravenous infusion of a donor's white blood cells collected after treatment with mobilization with filgrastim (G-CSF)
  Other Names: Allogeneic peripheral blood progenitor cell (PBPC) transplantation
Procedure: Total lymphoid irradiation (TLI) — TLI is administered in 80cGy fractions on Days -11 to Day-7 relative to allo-HSCT
Drug: Rituximab — 375 mg/m2 IV days 1 and 7 over 4 to 8 hours
  Other Names: Rituxan; Mabthera
Drug: Carmustine — Based on body weight, unless its more than 15 kg greater than the idal body 15mg/kg (max dose 550 mg/m2) day -6 over 2 hours.
  Males IBW = 50 kg + 2.3 kg/inch over 5 feet Females IBW = 45.5 kg + 2.3 kg/inch over 5 feet Adjusted IBW = IBW + 50% (actual weight - IBW)
  Other Names: BCNU; BiCNU
Drug: Etoposide — 60 mg/kg over 4 hours day -4 and alternatively VP-16 2 Gm/m² may be used (for mobilization)
  Other Names: Eposin; Etopophos; Vepesid; VP-16
Drug: Filgrastim — 10 µg/kg/day subcutaneous starting Day 9 until last day of apheresis. 5 ug/kg actual body weight per day will be started at Day +6 after allo-HCT until hematologic recovery
  Other Names: Granulocyte colony-stimulating factor (G-CSF, GCSF); Colony-stimulating factor 3 (CSF-3)
Drug: Anti-thymocyte globulin (ATG) — 1.5 mg/kg/day for 5 days
Drug: Cyclosporine — 5.0 mg/kg twice daily from day -3 until after day +56
  Other Names: Cyclosporin; CSP
Drug: Mycophenolate mofetil (MMF) — 250 mg (total) twice daily, oral
  15 mg/kg po on day 0, at 5-10 hours after mobilized PBPC infusion is complete. On day +1 MMF is taken at 15 mg/kg po b.i.d. (30 mg/kg/day) if transplantation was using a matched related donor and 15 mg/kg po t.i.d if from a matched unrelated donor or a one antigen mismatched donor.
  Other Names: CellCept
Drug: Cyclophosphamide — 100 mg/kg will be administered over 2 hours on day -2
  Other Names: Cytoxan; Neosar
Drug: Acetaminophen — Pre-medication for rituximab and PBPC infusion. Administered at 650 mg by mouth 1 hour prior to infusion
  Other Names: Tylenol
Drug: Diphenhydramine — Pre-medication for rituximab and PBPC infusion. Administered at 50 mg intravenous 1 hour prior to infusion
  Other Names: Benadryl
Drug: Hydrocortisone — Pre-medication for the PBPC infusion. Administered at 100 mg intravenous 1 hour prior to infusion
  Other Names: Cortef
Drug: Methylprednisolone — Anti-reaction medication for the ATG infusion. Administered at 1 mg/kg, Day-11 to Day-7
  Other Names: Solu-Medrol

SUMMARY:
The purpose of this study is to determine if double autologous then allogeneic hematopoietic cell transplant may offer an improved treatment option for patients with relapsed diffuse large B-cell lymphoma (DLBCL) who are not likely to be cured by the conventional transplantation regimen.

DETAILED DESCRIPTION:
This study tests a tandem transplant approach that starts with transplantation of the participant's own hematopoietic (blood) cells, eg, autologous hematopoietic cell transplant (auto-HCT) as preparation for an subsequent matched-donor allogeneic HCT (allo-HCT).

Participants will be have progenitor cells (stem cells) mobilized into the peripheral blood with rituximab, chemotherapy (cyclophosphamide or etoposide), and filgrastim (G-CSF); undergo apheresis to collect autologous peripheral blood stem cells (PBSC, aka hematopoietic cells); and be re-infused with ≥ 3 x 10e6 CD34+ cells/kg (auto-HCT). Subsequently, participants will receive therapeutic, non-myeloablative chemotherapy (carmustine + cyclophosphamide + etoposide), then transplant conditioning [total lymphoid irradiation (TLI) + anti-thymocyte globulin (ATG)] followed by ≥ 2 x 10e6 CD34+ cells/kg allogeneic PBSC obtained from a human leukocyte antigen (HLA)-matched or HLA single allele / antigen-mismatched donor (allo-HCT). Donors will be mobilized with 16 µg/kg filgrastim. Participant allo-HCT transplant is to occur within 150 days of auto-HCT. Post-allo-HCT infusion treatment includes cyclosporine and mycophenolate mofetil (MMF)

Subject's participation ends if a suitable matched donor is not identified within the 150 days.

Pre-medication treatments administered during this study may include acetaminophen; diphenhydramine; hydrocortisone; and methylprednisolone.

ELIGIBILITY:
INCLUSION CRITERIA

* Age 18 to 70 years.
* Histologically-proven diffuse large B-cell lymphoma (DLBCL) by the World Health Organization (WHO) classification.
* Relapse after achieving initial remission or failure to achieve initial remission. Patients with residual radiographic abnormalities after primary therapy are eligible if abnormalities are postive by fluorodeoxyglucose (FDG)-positron emission tomography (PET) (FDG-PET).
* Receipt of 2 cycles of second-line therapy and FDG-PET positive per Stanford (central) review. FDG-PET to be done 2 weeks after cycle 2 of second line chemotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status < 2
* Matched related or unrelated donor identified and available
* Bone marrow biopsy and cytogenetic analysis within 8 weeks of registration
* Pretreatment serum bilirubin < 2 x the institutional upper limit of normal (ULN)
* Serum creatinine < 2 x the institutional ULN and measured or estimated creatinine clearance > 60 mL/min by the following formula (all tests must be performed within 28 days prior to registration):

  * Estimated Creatinine Clearance = (140 age) x weight (kg) x 0.85 if female 72 x serum creatinine (mg/dL).
* EKG within 42 days prior to registration with no significant abnormalities suggestive of active cardiac disease
* Patients must have a radionuclide ejection fraction within 42 days of registration. If the ejection fraction is < 40%, the patient will not be eligible. If the ejection fraction is 40-50%, the patient will have a cardiology consult.
* Corrected diffusion capacity > 55%.
* Sexually active males are advised to use an accepted and effective method of birth control
* Women of child-bearing potential are advised to use an accepted and effective method of birth control
* Patients must sign and give written informed consent in accordance with institutional and federal guidelines. Patients must be informed of the investigational nature of this study.

EXCLUSION CRITERIA

* Known allergy to etoposide or a history of Grade 3 hemorrhagic cystitis with cyclophosphamide
* Greater than Grade 2 sensory or motor peripheral neuropathy from prior vinca alkaloid use
* Requiring therapy for coronary artery disease, cardiomyopathy, dysrhythmia, or congestive heart failure
* Known to be human immunodeficiency virus (HIV)-positive. The antibody test for HIV must be performed within 42 days of registration.
* Prior chemotherapy other than corticosteroids administered within 2 weeks of the initiation of protocol therapy.
* Prior malignancy, except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer or other cancer for which the patients has been disease-free for five years.
* Prior diagnosis of non-Hodgkin's lymphoma
* Active infection requiring oral or intravenous antibiotics
* Prior autologous or allogeneic hematopoietic cell transplantation
* Prior radioimmunotherapy
* Pregnant
* Lactating

DONOR ELIGIBILITY

* Related or unrelated HLA-identical donors who are in good health and have no contra-indication to donation
* No contra-indication for the donor to collection by apheresis of mononuclear cells mobilized by G-CSF at a dose of 16 µg/kg of body weight.
* Donors will be evaluated with a full history and physical examination.
* Virology testing including HIV; cytomegalovirus (CMV); Epstein-Barr virus (EBV); human T-lymphotropic virus (HTLV); rapid plasma reagin (RPR); Hepatitis A, B and C be performed within 30 days of donation.
* Prospective donors will be screened for CMV seroreactivity and seronegative donors will be utilized if available.
* If more than one human leukocyte antigen (HLA)-matched related donor exists, then the donor will be selected on the basis of CD31 allotype.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2006-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Kai Weng, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Autologous Peripheral Stem Cells
Arm/Group | Auto-HCT Followed by Allo-HCT for Poor-risk DLBCL
Started | 3
Completed | 3
Not Completed | 0
Period: Inter-treatment Period
Arm/Group | Auto-HCT Followed by Allo-HCT for Poor-risk DLBCL
Started | 3
Completed | 2
Not Completed | 1
Not completed — Disease progression | 1
Period: Allogeneic Peripheral Stem Cells
Arm/Group | Auto-HCT Followed by Allo-HCT for Poor-risk DLBCL
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Auto-HCT Followed by Allo-HCT for Poor-risk DLBCL
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS) Per Protocol
Description: Event-free survival (EFS) through 4 years, as assessed in participants with poor-risk recurrent or primary refractory DLBCL treated with TLI and ATG followed by matched allogeneic hematopoietic cell transplantation as a consolidation to HCT. Event is defined as tumor progression or death.
Time Frame: 48 months
Population: Reported data values are limited by protocol-specified upper boundary for the timeframe of this assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Auto-HCT Followed by Allo-HCT for Poor-risk DLBCL
Number analyzed (Participants) | 2
months | 48 [48 to 48]

2. Secondary Outcome: Median Time to Neutrophil Engraftment After Autologous Transplant
Description: Reported as neutrophil engraftment after autologous transplant, defined as absolute neutrophil count (ANC) > 500/µL, counting from the day of transplant.
Time Frame: within 1 month
Measure: Median (Full Range); unit: Days
Arm/Group | Auto-HCT Followed by Allo-HCT for Poor-risk DLBCL
Number analyzed (Participants) | 3
Days | 11 [9 to 12]

3. Secondary Outcome: Median Time to Platelet Engraftment After Autologous Transplant
Description: Reported as platelet engraftment after autologous transplant, defined as platelet count > 20,000/µL, counting from the day of transplant.
Time Frame: within 1 month
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Auto-HCT Followed by Allo-HCT for Poor-risk DLBCL
Number analyzed (Participants) | 3
Days | 19 [15 to 19]

4. Secondary Outcome: Median Time to Neutrophil Engraftment After Allogeneic Transplant
Description: Reported as neutrophil engraftment after allogeneic transplant, defined as absolute neutrophil count (ANC) > 500/µL, counting from the day of transplant.
Time Frame: within 1 month
Measure: Median (Full Range); unit: Days
Arm/Group | Auto-HCT Followed by Allo-HCT for Poor-risk DLBCL
Number analyzed (Participants) | 2
Days | 10.5 [9 to 12]

5. Secondary Outcome: Median Time to Platelet Engraftment After Allogeneic Transplant
Description: Reported as platelet engraftment after allogeneic transplant, defined as platelet count > 20,000/µL, counting from the day of transplant.
Time Frame: within 1 month
Population: Note: all participants engrafted platelets on the same day (see below for data values).
Measure: Median (Full Range); unit: Days
Arm/Group | Auto-HCT Followed by Allo-HCT for Poor-risk DLBCL
Number analyzed (Participants) | 2
Days | 10 [10 to 10]

6. Secondary Outcome: Incidence of Chronic Graft vs Host Disease (GvHD)
Description: The incidence of chronic graft vs host disease (GvHD) is reported as any events within 3 years. Note that GvHD was assessed per investigator judgement. There was no protocol-specified criteria of GvHD.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Auto-HCT Followed by Allo-HCT for Poor-risk DLBCL
Number analyzed (Participants) | 3
Participants | 0

7. Secondary Outcome: Overall Survival (OS)
Description: To evaluate the overall and transplant related mortality rate, reported as the number of subjects remaining alive 3 years after transplant.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Auto-HCT Followed by Allo-HCT for Poor-risk DLBCL
Number analyzed (Participants) | 3
Participants | 2

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Auto-HCT Followed by Allo-HCT for Poor-risk DLBCL
Serious Adverse Events (participants affected / at risk) | 3/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Auto-HCT Followed by Allo-HCT for Poor-risk DLBCL (N=3)
Platelet count decrease (Blood and lymphatic system disorders) | 1 (1)
Recurrent lymphoma (Blood and lymphatic system disorders) | 1 (2) — Includes progressive lymphoma
lymph nodes (Blood and lymphatic system disorders) | 1 (2) — left groin
Nausea (Gastrointestinal disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 2 (2)
Febrile neutropenia (Infections and infestations) | 2 (2)
Thrush (Skin and subcutaneous tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Auto-HCT Followed by Allo-HCT for Poor-risk DLBCL (N=3)
Bacteremia (Infections and infestations) | 1 (1)
facial cellulitis (Infections and infestations) | 1 (1)
Fever (Infections and infestations) | 3 (3) — Includes: Febrile Neutropenia
Headache (General disorders) | 1 (1)
Hypermetabolic lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) — In the necksupraclavicular area, axilla, chest wall, and groin.
Leukopenic (Blood and lymphatic system disorders) | 1 (1)
Maculo-papular rash (Skin and subcutaneous tissue disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Residual disease (Infections and infestations) | 1 (1) — in the left groin
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrush (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No